CLINICAL TRIAL: NCT06916884
Title: Confirmatory Study on the Efficacy and Safety of the Fixed-dose Combination of Desloratadine/Betamethasone Versus Desloratadine as Treatment in Patients With Allergic Rhinitis
Brief Title: Confirmatory Study on the Efficacy and Safety of the Fixed-dose Combination of Desloratadine/Betamethasone Versus Desloratadine
Acronym: DESCUBRA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30810-III-23(1)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Allergic Rhinitis
Keywords: rhinitis; allergies; respiratory system
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis; Hypersensitivity | interventions — desloratadine; Betamethasone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Desloratadine 5 mg + Betamethasone 0.25 mg (Experimental): Administered orally, one tablet a day, for 10 days.
  Interventions: Drug: Desloratadine / Betamethasone in fixed dose
- Group B: Desloratadine 5 mg (Active Comparator): Administered orally, one tablet a day, for 10 days.
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine / Betamethasone in fixed dose — 1 tablet, once a day of 5 mg / 0.25 mg
  Other Names: DESLORA / BETA
  Arms: Group A: Desloratadine 5 mg + Betamethasone 0.25 mg
Drug: Desloratadine — 1 tablet, once a day of 5 mg
  Other Names: DESLORA
  Arms: Group B: Desloratadine 5 mg

SUMMARY:
Phase IIIb , longitudinal, multicenter, randomized, double-blind, to evaluate efficacy and safety of the fixed-dose combination of Desloratadine 5 mg / Betamethasone 0.25 mg versus Desloratadine 5 mg monotherapy as treatment for symptoms associated with allergic rhinitis.

DETAILED DESCRIPTION:
Nasal symptom changes will be assessed daily over a 10-day intervention period using the Total Nasal Symptom Score (TNSS) for allergic rhinitis. Patients will complete the first questionnaire during the randomization visit, followed by daily entries each night before bedtime using a patient diary. The final assessment will be completed during the study's end-of-treatment visit.

Quality of life, global clinical impression, and patient global assessment will be evaluated during in-person visits conducted at baseline, Day 5, and Day 10.

The incidence of adverse events throughout the study will be analyzed by treatment group and reported as frequencies and percentages. Events will be classified according to frequency, seriousness, severity, and their relationship to the investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and able to provide written informed consent.
* Clinical diagnosis (based on medical history and physical examination) of active allergic rhinitis at study entry.
* Patients presenting with moderate to severe nasal symptoms, with a Total Nasal Symptom Score (TNSS) ≥5.
* In the case of women of childbearing potential who are sexually active, the use of an acceptable contraceptive method (barrier and/or hormonal), as determined by the investigator.
* In the opinion of the Principal Investigator or treating physician, the patient is indicated for treatment with the investigational product and may derive clinical benefit from it.

Exclusion Criteria:

* Patients for whom the investigational drug is medically contraindicated.
* Known allergy or hypersensitivity to the active ingredient, study medications, related products, or excipients.
* History of nasal trauma (surgical or accidental) within the past week.
* Positive pregnancy test, pregnant or breastfeeding women, or women planning to become pregnant during the course of the study.
* Acute or chronic lower or upper respiratory tract infections, such as the common cold, influenza, pneumonia, bronchitis, or chronic sinusitis.
* History of non-allergic rhinitis, such as chronic non-allergic rhinitis, drug-induced rhinitis, atrophic rhinitis, hormonal rhinitis, or unilateral rhinitis, as reported in the medical history or patient interview.
* History of nasal polyposis, primary ciliary dyskinesia syndrome, and/or non-allergic rhinitis with eosinophilia syndrome (NARES).
* Current smokers, or history of alcohol and/or drug abuse in the past year according to DSM-V criteria.
* History of seizure disorders, status epilepticus, or generalized tonic-clonic seizures.
* History of chronic hepatic failure classified as Child-Pugh C, as reported in the medical history or patient interview.
* History of chronic renal failure (glomerular filtration rate < 30 mL/min/1.73 m²), as reported in the medical history or patient interview.
* Any condition, in the investigator's opinion, that affects prognosis or precludes outpatient management, which must be evaluated by the principal investigator to determine the subject's eligibility.
* History of severe, progressive, unstable, or advanced disease of any kind that could interfere with efficacy and safety evaluations or pose a risk to the patient.
* Oncology patients (except those with basal cell skin cancer) or patients with serious illnesses who, in the investigator's opinion, have a poor prognosis or life expectancy of less than one year, including those with mental health disorders.
* Active participation in another clinical trial involving an investigational treatment or participation in any clinical study within the previous two weeks.
* Patients whose participation in the study may be influenced (e.g., employees of the research center or sponsor, incarcerated individuals, etc.).
* Patients with symptoms suggestive of active COVID-19 infection (e.g., fever, cough, dyspnea) and/or contact within the past 14 days with a suspected or confirmed COVID-19 case and/or a positive COVID-19 test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-05-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of the magnitude of change in the TNSS over the 10-day intervention period versus the baseline, by treatment group. | 10 days
  The Total Nasal Symptom Score (TNSS) is a clinical measure used to assess the severity of nasal symptoms in patients, particularly those suffering from allergic rhinitis. It assess the four cardinal symptoms of allergic rhinitis: sneezing, rhinorrhea (nasal mucus discharge), nasal pruritus (itching), and nasal obstruction (difficulty breathing). According to the evaluation the magnitude of the symptoms could be classified as: None, Mild, Moderate and Severe.
  The researcher will apply the TNSS score to each patient at each visit and follow up call, to assess improvement in symptoms. At the end of the clinical trial the magnitude of change will be measured and compared between treatment groups.
will be measured and compared between treatment groups. | 10 days
  To describe the frequency, intensity and causality of the adverse events presented during the clinical trial by treatment group. The adverse events will be registered by the patient in the diary record. Each adverse event will be followed up at the discretion of the researcher.

SECONDARY OUTCOMES:
Compare quality of life, measured as the change in score on the modified Likert scale for this outcome, by treatment group, at days 5 and 10 of the intervention compared to baseline. | 10 days
  A Likert scale for quality of life is a rating scale used to measure opinions, attitudes, or behaviors. It consists of a statement or a question, followed by a series of six answer statements. Quality of life should be assessed by the principal investigator or designated physician at each visit.
Describe disease severity and improvement using the CGI scale by treatment group, at days 5 and 10 of the intervention compared to baseline. | 10 days
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. The evaluation range goes from 1 - 7: 1- Marked improvement, 2- improvement, 3- slightly improved, 4- no change, 5- slightly worsened, 6- worsened, and 7- markedly worsened.
Describe the PGA of the treatment received at days 5 and 10 of the intervention, by treatment group. | 10 days
  Patient's Global Assessment (PGA) is often assessed by a single question with a 0-4 response. On Days 5 and 10 of the intervention, a PGA of response to treatment will be conducted, using a scoring scale from 0 to 4, with 4 representing the worst possible assessment.

OTHER OUTCOMES:
To report the percentage of therapeutic adherence at day 10 of the intervention in each treatment group. | 10 days
  Therapeutic adherence will be defined by the principal researcher. Adherence to treatment will be defined as a consumption ≥ 80% of the doses that the patient should have ingested at the time of the corresponding evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Murguía Martín, MD, Principal Investigator — Unidad de Medicina Especializada SMA; Tobías Avendaño Santiago, MD, Principal Investigator — Oaxaca Site Management Organization, S.C; Erika N Durón López, MD, Principal Investigator — Centro de Investigación Médica de Aguascalientes; María D Escobar Zalapa, MD, Principal Investigator — CICMEX Centro de Investigación Clínica de México S de RL de CV
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] RICKHAM PP. HUMAN EXPERIMENTATION. CODE OF ETHICS OF THE WORLD MEDICAL ASSOCIATION. DECLARATION OF HELSINKI. Br Med J. 1964 Jul 18;2(5402):177. doi: 10.1136/bmj.2.5402.177. No abstract available. PMID 14150898
- [Background] Shukla AK, Jhaj R, Misra S, Ahmed SN, Nanda M, Chaudhary D. Agreement between WHO-UMC causality scale and the Naranjo algorithm for causality assessment of adverse drug reactions. J Family Med Prim Care. 2021 Sep;10(9):3303-3308. doi: 10.4103/jfmpc.jfmpc_831_21. Epub 2021 Sep 30. PMID 34760748
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Comite Nacional de Endocrinologia. [Considerations for safe glucocorticoid therapy]. Arch Argent Pediatr. 2018 Jun 1;116(3):s71-s76. doi: 10.5546/aap.2018.s71. Spanish. PMID 35786822
- [Background] Horak F, Stubner UP, Zieglmayer R, Harris AG. Effect of desloratadine versus placebo on nasal airflow and subjective measures of nasal obstruction in subjects with grass pollen-induced allergic rhinitis in an allergen-exposure unit. J Allergy Clin Immunol. 2002 Jun;109(6):956-61. doi: 10.1067/mai.2002.124657. PMID 12063524
- [Background] Simons FE, Prenner BM, Finn A Jr; Desloratadine Study Group. Efficacy and safety of desloratadine in the treatment of perennial allergic rhinitis. J Allergy Clin Immunol. 2003 Mar;111(3):617-22. doi: 10.1067/mai.2003.168. PMID 12642846
- [Background] Mendoza de Morales T, Sanchez F. Clinical efficacy and safety of a combined loratadine-betamethasone oral solution in the treatment of severe pediatric perennial allergic rhinitis. World Allergy Organ J. 2009 Apr;2(4):49-53. doi: 10.1097/WOX.0b013e31819f2105. PMID 23282980
- [Background] Wandalsen GF, Miranda C, Ensina LF, Sano F, Amazonas RB, Silva JMD, Sole D. Association between desloratadine and prednisolone in the treatment of children with acute symptoms of allergic rhinitis: a double-blind, randomized and controlled clinical trial. Braz J Otorhinolaryngol. 2017 Nov-Dec;83(6):633-639. doi: 10.1016/j.bjorl.2016.08.009. Epub 2016 Sep 13. PMID 27670203
- [Background] Murdoch D, Goa KL, Keam SJ. Desloratadine: an update of its efficacy in the management of allergic disorders. Drugs. 2003;63(19):2051-77. doi: 10.2165/00003495-200363190-00010. PMID 12962522
- [Background] Bachert C. A review of the efficacy of desloratadine, fexofenadine, and levocetirizine in the treatment of nasal congestion in patients with allergic rhinitis. Clin Ther. 2009 May;31(5):921-44. doi: 10.1016/j.clinthera.2009.05.017. PMID 19539095
- [Background] Snyman JR, Potter PC, Groenewald M, Levin J; Claricort Study Group. Effect of betamethasone-loratadine combination therapy on severe exacerbations of allergic rhinitis : a randomised, controlled trial. Clin Drug Investig. 2004;24(5):265-74. doi: 10.2165/00044011-200424050-00003. PMID 17503888
- [Background] Bernstein DI, Schwartz G, Bernstein JA. Allergic Rhinitis: Mechanisms and Treatment. Immunol Allergy Clin North Am. 2016 May;36(2):261-78. doi: 10.1016/j.iac.2015.12.004. Epub 2016 Mar 10. PMID 27083101
- [Background] May JR, Dolen WK. Management of Allergic Rhinitis: A Review for the Community Pharmacist. Clin Ther. 2017 Dec;39(12):2410-2419. doi: 10.1016/j.clinthera.2017.10.006. Epub 2017 Oct 25. PMID 29079387
- [Background] Eifan AO, Durham SR. Pathogenesis of rhinitis. Clin Exp Allergy. 2016 Sep;46(9):1139-51. doi: 10.1111/cea.12780. PMID 27434218
- [Background] Greiner AN, Hellings PW, Rotiroti G, Scadding GK. Allergic rhinitis. Lancet. 2011 Dec 17;378(9809):2112-22. doi: 10.1016/S0140-6736(11)60130-X. Epub 2011 Jul 23. PMID 21783242
- [Background] Meltzer EO, Rosario NA, Van Bever H, Lucio L. Fexofenadine: review of safety, efficacy and unmet needs in children with allergic rhinitis. Allergy Asthma Clin Immunol. 2021 Nov 2;17(1):113. doi: 10.1186/s13223-021-00614-6. PMID 34727966